CLINICAL TRIAL: NCT05856097
Title: Effects of Kinesio Taping With and Without Diaphragmatic Breathing on Incisional Pain and Mobility in Women After Cesarean Section
Brief Title: Kinesio Taping With and Without Diaphragmatic Breathing in Women After Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0519
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Cesarean Section Complications
Keywords: Ache; Breathing Exercises
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesio taping with diaphragmatic breathing (Experimental): kinesio taping application with diaphragmatic breathing
  Interventions: Other: kinesio taping with diaphragmatic breathing
- kinesio taping without diaphragmatic breathing (Active Comparator): kinesio taping application without diaphragmatic breathing
  Interventions: Other: kinesio taping without diaphragmatic breathing

INTERVENTIONS:
Other: kinesio taping with diaphragmatic breathing — .kinesio tape was applied on1st day of intervention with the 20 minutes session of diaphragmatic breathing 3 sessions were given
  Arms: kinesio taping with diaphragmatic breathing
Other: kinesio taping without diaphragmatic breathing — kinesio tape was applied day 1st of intervention. 3 sessions were given
  Arms: kinesio taping without diaphragmatic breathing

SUMMARY:
Cesarean section is a major abdominal surgery and major challenge of it is to manage the pain and make the patient mobile .In spite of the advantageous effects of kinesio taping and diaphragmatic breathing, limited, data reported to study analgesic effects on pain management and mobility restoration in acute phase of cesarean section.. This study will aim to meet the dares which are associated with cesarean section by reducing the incisional pain associated with improvement in physical mobility as a non-pharmacological treatment.

DETAILED DESCRIPTION:
In year 2022 conducted a study to evaluate the effects of kinesio taping with the breathing exercises on the management of pain after c section .Their title of study was The effects of Kinesio taping and breathing exercises on pain management after gynaecological abdominal surgery: A randomized controlled study. This study was conducted among 132 participants between June 2017 and 18.kinesio taping was applied immediately after the surgery and on the post op day 1, 2, 3 breathing exercises were performed for 30 mins three times a day. Their study concluded that kinesio taping is a reliable method to cover up the acute pain in the gynaecological abdominal surgery.

In the year 2022 a study was conducted with the title The effects of kinesio tape on low back pain and disability in pregnant women to scrutinize the effects of kinesio taping on low back pain and disability in pregnant females. It was a single blind clinical trial including 80 pregnant females. Two randomly assigned groups were made of in which pain was assessed by VAS before and after application of kinesio taping on the day 1st,2nd,7th,and 14th. Disability was measured by Roland-Morris disability questionnaire before and after intervention on day 7th and 14th. Their result concludes that kinesio taping have lasting effects on low back pain disability and reduced disability was noticed .In the year 2020 another study was conducted to study the effects of KT on the pain, anxiety, menstrual cramps in the women with primary dysmenorrhea with the comparison with control and sham tape.51 women with the PD were categorized in the three groups KT, sham tape and control group. KT was applied at the sacral and supra pubic region with the ligament technique in KT group and applied on the trochanter major with no technique in the sham tape group. Pain, anxiety level, and menstrual complaints were examined before and after intervention. Their was positive response of the study responding to the decrease in anxiety level menstrual cramps and pain.

To the best of researchers knowledge, there is not enough literature present which can justify the efficacy of these interventions in a justified manner. Data is not sufficient that supports combined efficacy of these two interventions after cesarean section regarding pain management and mobility.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous patients
* Participants having no serious medical illness

Exclusion Criteria:

* Multi gravida patients
* Any serious morbidity
* Patient gone through any other abdominal surgery except of cesarean section
* Patients with the infectious wound

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females are included for the study to record the results after cesarean birth process.
Enrollment: 36 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-09-03 (Estimated); Study Completion 2023-10-03 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | 4th week
  Changes from baseline A Visual Analogue Scale (VAS) is one of the pain rating scales used for the first time in 1921 by Hayes and Patterson. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. For example, the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Ask the patient to rate their current level of pain by placing a mark on the line.
bedside mobility assessment tool (BMAT) | 4th week
  Changes from baseline BMAT is a tool designed for nurses to assess patient mobility in acute care. The BMAT allows nurses (and other healthcare workers) to determine the appropriate patient handling and mobility equipment or device to safely move or mobilize the patient. It consists of four steps, first is sit and shake, second is stretch and point ,third is stand and fourth is step. Mobility level 1,2,3and 4 is given to patients according to their level of mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Mehjabeen, Principal Investigator — Riphah International University
Locations (1):
- District head quarter hospital jhang, Jhang, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WHO Recommendations Non-Clinical Interventions to Reduce Unnecessary Caesarean Sections. Geneva: World Health Organization; 2018. Available from http://www.ncbi.nlm.nih.gov/books/NBK532672/ PMID 30398818
- [Background] Weckesser A, Farmer N, Dam R, Wilson A, Morton VH, Morris RK. Women's perspectives on caesarean section recovery, infection and the PREPS trial: a qualitative pilot study. BMC Pregnancy Childbirth. 2019 Jul 15;19(1):245. doi: 10.1186/s12884-019-2402-8. PMID 31307417
- [Background] Singla N, Garg K, Jain R, Malhotra A, Singh MR, Grewal A. Analgesic efficacy of dexamethasone versus dexmedetomidine as an adjuvant to ropivacaine in ultrasound-guided transversus abdominis plane block for post-operative pain relief in caesarean section: A prospective randomised controlled study. Indian J Anaesth. 2021 Sep;65(Suppl 3):S121-S126. doi: 10.4103/ija.IJA_228_21. Epub 2021 Sep 15. PMID 34703057
- [Background] Toprak Celenay S, Kavalci B, Karakus A, Alkan A. Effects of kinesio tape application on pain, anxiety, and menstrual complaints in women with primary dysmenorrhea: A randomized sham-controlled trial. Complement Ther Clin Pract. 2020 May;39:101148. doi: 10.1016/j.ctcp.2020.101148. Epub 2020 Mar 18. PMID 32379680
- [Background] Aalishahi T, Maryam-Lotfipur-Rafsanjani S, Ghorashi Z, Sayadi AR. The Effects of Kinesio Tape on Low Back Pain and Disability in Pregnant Women. Iran J Nurs Midwifery Res. 2022 Jan 25;27(1):41-46. doi: 10.4103/ijnmr.IJNMR_291_20. eCollection 2022 Jan-Feb. PMID 35280198
- [Background] Shahbazi M, Sarrafzadeh J, Fatemi TS, Hafizi L. Effect of thoracic Kinesio taping on acute lumbar and leg pain in a pregnant woman: A case report. Sports Orthopaedics and Traumatology. 2021.
- [Background] Espi-Lopez GV, Ingles M, Ferrando AC, Serra-Ano P. Effect of Kinesio taping on clinical symptoms in people with fibromyalgia: A randomized clinical trial. J Back Musculoskelet Rehabil. 2019;32(4):561-567. doi: 10.3233/BMR-171100. PMID 30530959
- [Background] Yilmaz S, Terzioglu F. The effects of Kinesio taping and breathing exercises on pain management after gynaecological abdominal surgery: A randomized controlled study. Int J Nurs Pract. 2023 Apr;29(2):e13088. doi: 10.1111/ijn.13088. Epub 2022 Aug 4. PMID 35929048
- [Background] Hamasaki H. Effects of Diaphragmatic Breathing on Health: A Narrative Review. Medicines (Basel). 2020 Oct 15;7(10):65. doi: 10.3390/medicines7100065. PMID 33076360
- [Background] Kuravskaya YV, Aravitskaya M. EFFECTIVENESS OF RECOVERY OF THE PSYCHO-EMOTIONAL AND PHYSICAL STATUS OF WOMEN WHO HAVE SUFFERED A CAESAREAN SECTION BY MEANS OF PHYSICAL THERAPY. Art of Medicine. 2022:50-5.
- [Background] Mohamed H, Yousef A, Kamel H-E, Oweda K, Abdelsameaa G. Kinesio Taping and Strength Recovery of Postnatal Abdominal Muscles after Cesarean Section. Egyptian Journal of Physical Therapy. 2020;4(1):13-9.
- [Background] Nugent SM, Lovejoy TI, Shull S, Dobscha SK, Morasco BJ. Associations of Pain Numeric Rating Scale Scores Collected during Usual Care with Research Administered Patient Reported Pain Outcomes. Pain Med. 2021 Oct 8;22(10):2235-2241. doi: 10.1093/pm/pnab110. PMID 33749760
- [Background] Rose A, Carter N, Vann C, Lloyd-Penza M, Andrusko M. Implementing Bedside Mobility Assessment Tool to Improve Patient Outcomes and Staff Communication. Medsurg Nursing. 2022;31(1):32-6.
- [Background] Boynton T, Kumpar D, VanGilder C. The bedside mobility assessment tool 2.0. American Nurse Journal. 2020;15(7):15.